CLINICAL TRIAL: NCT03999437
Title: EFFICACY AND SAFETY OF A SINGLE-APPLICATION TREATMENT USING TERBINAFINE HYDROCHLORIDE (1%) TOPICAL LIQUID SOLUTION VERSUS A SINGLE-APPLICATION TREATMENT USING BUTENAFINE HYDROCHLORIDE (1%) TOPICAL LIQUID SOLUTION FOR THE TREATMENT OF TINEA PEDIS: A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED TRIAL
Brief Title: SINGLE-APPLICATION TERBINAFINE HYDROCHLORIDE (1%) TOPICAL LIQUID SOLUTION VERSUS A SINGLE-APPLICATION BUTENAFINE HYDROCHLORIDE (1%) TOPICAL LIQUID SOLUTION FOR THE TREATMENT OF TINEA PEDIS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: United Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RD2018-02
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis | interventions — Terbinafine; butenafine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment # 1 (Experimental)
  Interventions: Drug: TERBINAFINE HYDROCHLORIDE (1%)
- Treatment # 2 (Experimental)
  Interventions: Drug: BUTENAFINE HYDROCHLORIDE (1%)
- Placebo Control (Placebo Comparator)
  Interventions: Drug: Vehicle Control

INTERVENTIONS:
Drug: TERBINAFINE HYDROCHLORIDE (1%) — Topical liquid solution
  Arms: Treatment # 1
Drug: BUTENAFINE HYDROCHLORIDE (1%) — Topical liquid solution
  Arms: Treatment # 2
Drug: Vehicle Control — Topical liquid solution
  Arms: Placebo Control

SUMMARY:
Tinea pedis or athlete's foot is the most common fungal infection worldwide, caused by infection of the feet with dermatophytes such as Trichophyton rubrum, Trichophyton interdigitale (formerly Trichophyton mentagrophytes), and Epidermophyton floccosum. Diagnosis of tinea pedia involves clinical symptoms as well as microscopic examination. Topical therapies are usually applied once or twice daily for as long as 4 weeks, posing a challenge to compliance. The current study aims to test a formulation of the single-dose 1% terbinafine hydrochloride, as well as a single-dose 1% butenafine hydrochloride, versus a vehicle control in adult Filipino patients with athlete's foot. This study will benefit the Filipino community by helping us determine which anti-fungal cream is most effective for athlete's foot.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant females aged 18-60 years old.
* Clinical diagnosis of tinea pedis (total sign/symptom score >2), lesions between the toes, with possible extension to the lateral surfaces and soles of the feet confirmed by a positive microscopy prior to dosing.
* Willing to sign the informed consent.

Exclusion Criteria:

* Females who are pregnant (confirmed by a pregnancy test), suspect themselves to be pregnant (even if pregnancy test is negative), breast-feeding, or planning a pregnancy.
* Signs of systemic or other superficial fungal disease (e.g.onychomycosis), clinically relevant abnormal findings upon physical examination of the foot or previous treatment with a disallowed medication (such as corticosteroids).
* Presence of non-healing wounds and/or bacterial infection on the feet.
* Secondary bacterial infection due to tinea pedis
* Presence of pigmentation, extensive scarring, or pigmented lesions in the treatment areas, which could interfere with the rating of efficacy parameters.
* History of hypersensitivity to any component of the test products.
* Current imuunosuppression. Specifically, these include ￼patients with co-morbidities such as diabetes, HIV, chronic diseases requiring maintenance medications, acute febrile/infectious illnesses (i.e. Dengue, pneumonia, etc)
* Use within 3 months prior to baseline of: 1.) chemotherapy, or 2.) radiation therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-12-13 (Estimated); Study Completion 2020-01-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with effective treatment at week 6 | 6 weeks
  Defined as negative microscopy and improvement in signs and symptoms: mild or no erythema, desquamation or pruritis (<=1), no vesiculation, and a total sign/symptom score of <=2.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Management and Testing Associates, Inc., City of Muntinlupa, Philippines